CLINICAL TRIAL: NCT04175587
Title: Implement Randomized, Controlled, International Multi-center Clinical Trial of Compound Realgar-Indigo Naturalis Formula Plus Retinoic Acid for Non-high-risk Acute Promyelocytic Leukaemia
Brief Title: Randomized,International Multi-center Clinical Trial of RIF Plus RA for Non-high-risk APL
Acronym: RIF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, Xiaojun Huang,MD, Director of Hematology Department, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RIF & ATRA in NHR APL
Record Dates: First submitted 2019-11-21; First posted 2019-11-25 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Acute Promyelocytic Leukaemia
Keywords: Realgar-Indigo Naturalis Formula, Retinoic Acid
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Tretinoin

STUDY DESIGN:
Intervention Model Description: This study is a prospective, non-inferiority, randomized controlled clinical trial. The non-inferiority is concluded if the lower limit of the 95% CI for the difference in proportion of patients achieving EFS is greater than the -10% non-inferiority margin. The survival curves are estimated by using the Kaplan-Meier method and will be compared by using the log-rank test.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compound Realgar-Indigo Naturalis Formula Plus Retinoic Acid (Experimental): Induction: a) RIF: 60 mg/kg daily until CR, b) ATRA: 25 mg/m² daily until CR; Consolidation: a) RIF: 60 mg/kg daily, in a 4-week on 4-week off regimen for four cycles in a 4-week on 4-week off regimen for four cycles b) ATRA: 25 mg/m² daily, in a 2-week on 2-week off regimen for seven cycles
  Interventions: Drug: Compound Realgar-Indigo Naturalis Formula Plus Retinoic Acid
- Arsenic trioxide Plus Retinoic Acid (Other): Induction: a) Arsenic trioxide: 0·15 mg/kg daily until CR, b) ATRA: 25 mg/m² daily until CR Consolidation: a) Arsenic trioxide: 0.15mg/kg daily, in a 4-week on 4-week off regimen for four cycles b) ATRA: 25 mg/m² daily, in a 2-week on 2-week off regimen for seven cycles Expected Efficacy: Oral RIF plus ATRA is not inferior to intravenous arsenic trioxide plus ATRA for achieving 2-year EFS.
  Interventions: Drug: Compound Realgar-Indigo Naturalis Formula Plus Retinoic Acid

INTERVENTIONS:
Drug: Compound Realgar-Indigo Naturalis Formula Plus Retinoic Acid — Randomization is done centrally according to trial centers Eligible patients are randomly assigned (2:1) to the Treatment Group or the Control Group, with a 24-month follow-up.
  Other Names: intravenous arsenic trioxide plus Retinoic Acid

SUMMARY:
Acute Promyelocytic Leukaemia (APL) has been known as a type of cancer, which is of great significance to improve its eradication rate. Recent clinical trials show that ATRA plus ATO treatment regimen can result in complete response (CR) in 90-94% of patients and 5-year disease-free survival (DFS) in more than 90% of patients. However, the ATRA plus ATO treatment regimen can achieve considerate survival rate, patients still need to receive infusion therapy in hospital. If oral arsenic can replace intravenous ATO without reduction of the efficacy, patients would not need to be administered to receive treatment, which would highly increase their quality of lives. Phase I, II Clinical trials have verified the security and efficacy of the Compound Realgar-Indigo Naturalis Formula. Compound Realgar-Indigo Naturalis Formula was approved by the China Food and Drug Administration in 2009. Investergators have done a multi-centre, randomized, controlled, non-inferiority phase 3 clinical trial in China. And the result showed that oral arsenic plus retinoic acid has an anti-leukaemic efficacy similar to the intravenous arsenic treatment. So Investigators performed an international multi-center, Randomized controlled clinical trialsto compare the efficacy of oral RIF plus ATRA with intravenous arsenic trioxide plus ATRA in patients with non-high-risk APL in different racial types.

DETAILED DESCRIPTION:
Acute Promyelocytic Leukaemia (APL) has been known as a type of cancer, seriously endangering human health especially for young adults. It is of great significance to improve its eradication rate. Recent clinical trials show that ATRA plus ATO treatment regimen can result in complete response (CR) in 90-94% of patients and 5-year disease-free survival (DFS) in more than 90% of patients.

However, the ATRA plus ATO treatment regimen can achieve considerate survival rate, patients still need to receive infusion therapy in hospital. If oral arsenic can replace intravenous ATO without reduction of the efficacy, patients would not need to be administered to receive treatment, which would highly increase their quality of lives. The research and development of oral arsenic has therefore become a hotpoint. Professor Huang, Shilin from he 210th Hospital of PLA, according to the Prescription Theory "Jun Chen Zuo Shi", developed and designed an oral arsenic, the Compound Realgar-Indigo Naturalis Formula. Phase I, II Clinical trials have verified the security and efficacy of the Compound Realgar-Indigo Naturalis Formula. Research Team led by Professor Huang, Saijun, Shanghai Institute of Haematology (China), studied Compound Realgar-Indigo Naturalis Formula's mechanism of action from vitro cell lines and mice.

In the following Phase II clinical trial, APL patients received Compound Realgar-Indigo Naturalis Formula solo treatment regime. It resulted in 96.7% of CR and high safety rate Compound Realgar-Indigo Naturalis Formula was approved by the China Food and Drug Administration in 2009. Investigators have done a multi-centre, randomized, controlled, non-inferiority phase 3 clinical trial in China. 242 newly diagnosed APL patients (with newly diagnosed WBC<50×10^9/L) were enrolled. And the result showed that oral arsenic plus retinoic acid has an anti-leukaemic efficacy similar to the intravenous arsenic treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed APL patient (with WHO performance status)
2. Age 18-70
3. ALT and AST of maximum 2·5 times the ULN, and bilirubin concentration of maximum two times the ULN
4. Creatinine concentration of maximum three times the ULN
5. Performance status of 0-2 grade (ECOG)
6. WBC ≤ 10 x 109/L before the treatment
7. Informed Consent Paper signed

Exclusion Criteria:

1. Cerebral hemorrhage
2. Pregnancy
3. Concomitant severe psychiatric condition or anything else against the fulfillment of the plan
4. Clinically significant arrhythmias or electrocardiogram abnormalities (QT>500ms)
5. Refusal to sign off the Informed Consent Paper

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
2-year Event-free Survival (EFS) rate | 2 year after diagnosis
  treatment failure (no CR after 45-day induction therapy, or no molecular complete remission after 3-month consolidation therapy), relapse (molecular relapse, or haematological relapse); or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jun Huang, MD, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No